CLINICAL TRIAL: NCT01630876
Title: Anatomic and Functional Outcomes of 23-gauge Vitrectomy Combined With Posterior Subtenon Triamcinolone Injection for the Treatment of Idiopathic Epiretinal Membrane
Brief Title: Outcomes of Vitrectomy Combined With Subtenon Triamcinolone Injection for the Idiopathic Epiretinal Membrane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Min Sagong, Assistant Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YUH-12-0309-M2
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Epiretinal Membrane
Keywords: Epiretinal membrane; triamcinolone acetonide
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitrectomy only group (Sham Comparator): The patients who will underwent 23- gauge transconjunctival sutureless vitrectomy only.
  Interventions: Procedure: Vitrectomy only group
- Combined therapy group (Experimental): The patients who will underwent 23- gauge transconjunctival sutureless vitrectomy with concomitant posterior subtenon Triamcinolone acetate injection.
  Interventions: Procedure: Combined therapy group

INTERVENTIONS:
Procedure: Vitrectomy only group — The patients who will underwent 23- gauge transconjunctival sutureless vitrectomy only. The procedure will be done under retrobulbar anesthesia.
  Arms: Vitrectomy only group
Procedure: Combined therapy group — The patients who will underwent 23- gauge transconjunctival sutureless vitrectomy with concomitant posterior subtenon Triamcinolone acetate injection. For the posterior subtenon Triamcinolone acetate injection injection, a 1 ml of a 40 mg/ml of triamcinolone acetonide was given in the inferotemporal quadrant using a 27-gauge needle on 3-ml syringe. The conjunctiva and the Tenon's capsule were penetrated with the bevel of the needle toward the globe. The needle was advanced toward the macular area, taking care to remain in contact with the globe until the hub was firmly pressed against the conjunctival fornix and then the corticosteroid was slowly injected.
  Arms: Combined therapy group

SUMMARY:
This study compares the anatomical and visual outcomes of patients with idiopathic epiretinal membrane(ERM) treated by vitrectomy and membrane peeling with or without subtenon triamcinolone acetonide injection

ELIGIBILITY:
Inclusion Criteria:

* 1.The participant must have idiopathic epiretinal membrane 2.The participant must be willing and able to comply with the protocol.

Exclusion Criteria:

* 1. The participant has idiopathic epiretinal membrane with other ocular vascular diseases such as Diabetes retinopathy, BRVO, etc.

  2. The participant has any additional ocular diseases that have irreversibly compromised or could likely compromise the visual acuity of the study eye including amblyopia, anterior ischemic optic neuropathy, clinically significant diabetic macular edema, severe non proliferative diabetic retinopathy, or proliferative diabetic retinopathy.

  3. The participant has had intraocular surgery (including lens replacement surgery).

  4. The participant has a history of (within the last six months), or current ocular or periocular infection (including any history of ocular herpes zoster or simplex).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Changes of best corrected visual acuity and central retinal thickness | 6 months
  Changes of best corrected visual acuity and central retinal thickness on optical coherence tomography (OCT) at baseline and 1, 3, 6 months after injection

SECONDARY OUTCOMES:
Changes in status of ISOS line | 6 months
  Changes in status of ISOS line on optical coherence tomography (OCT) at baseline and 1, 3, 6 months after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam University College of Medicine, Daegu, South Korea